CLINICAL TRIAL: NCT05467007
Title: Urgent Care Management of Respiratory Illness Enabled With Novel Testing Pathway (URGENT): A Randomized Control Trial of Respiratory PCR Versus Standard Care
Brief Title: Urgent Care Management of Respiratory Illness Enabled With Novel Testing Pathway
Acronym: URGENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Meltzer (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor-Investigator, Andrew Meltzer, Chief, Clinical Research Section, Department of Emergency Medicine, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NCR213901
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Viral Infection; Acute Respiratory Infection; Upper Resp Tract Infection
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: 1 to 1 RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BioFire® Respiratory Panel 2.1-EZ (Experimental): EXP group will receive the BioFire RP2.1-EZ panel, designed to test for a variety of bacterial and/or viral causes for illness
  Interventions: Diagnostic Test: BioFire® Respiratory Panel 2.1-EZ
- Standard of Care (No Intervention): Standard care procedures are essentially yes/no to patient having SARS-COV-2, the SC group will receive the standard nasal swab used in the IPCs.

INTERVENTIONS:
Diagnostic Test: BioFire® Respiratory Panel 2.1-EZ — BioFire RP2.1-EZ Panel uses a syndromic approach to quickly identify SARS-CoV-2, along with 18 additional viral and bacterial pathogens in patients suspected of SARS-CoV-2. This PCR test provides results in about 45 minutes.
  Arms: BioFire® Respiratory Panel 2.1-EZ

SUMMARY:
Rapid diagnosis and precise treatment have become possible with multiplex polymerase chain reaction (PCR) panels that can identify a variety of causative agents of acute respiratory illnesses such as bacterial and viral infections in one urgent care visit. While real-time PCR is currently used as a standard for diagnosing acute respiratory illnesses such as influenza due to its high sensitivity and specificity, it typically takes several hours for results which is unfavorable in the urgent care setting. Highly sensitive and rapid random-access PCR tests provide the sensitivity and specificity needed to both rapidly and accurately diagnose acute respiratory illnesses. Similar PCR panels have been used in previous research for the diagnosis of gastrointestinal illnesses in the emergency department and point-of-care testing for hospitalized adults presenting with acute respiratory illness. In this study, the investigators aim to determine if a rapid multiplex PCR test for urgent care patients with symptomatic upper respiratory infections can improve patient and provider-reported outcomes. This study utilizes the Biofire® FilmArray Panel (RP2.1-EZ) which in previous studies has been shown to be highly effective in diagnosing acute respiratory illnesses.

DETAILED DESCRIPTION:
Research assistants in the IPCs will screen for possible participants by searching the electronic health record for complaints and/or symptoms of respiratory illness. Patients who screen eligible will be approached about potential interest, review inclusion and exclusion criteria, and obtain informed consent. All consented patients will be given a study ID and recorded in enrollment log. Patients who consent will be randomized to one of the two groups: BioFire® Respiratory Panel 2.1-EZ (RP2.1-EZ; EXP) versus standard care (SC). The RP2.1-EZ panel is designed to test for a variety of bacterial and/or viral causes for illness whereas standard care procedures are essentially yes/no to patient having SARS-COV-2. Both groups will receive a nasal swab, however, the EXP group will receive the BioFire RP2.1-EZ panel, and the SC group will receive the standard nasal swab used in the IPCs. As the RP2.1-EZ panel includes SARS-COV-2, patients in the EXP group need not receive two separate nasal swabs. Nasal swabs will be performed for both groups, ideally during triage, however, the sample may be collected any time during the visit, by staff trained by BioFire Diagnostics LLC. After the nasal swab is collected, it will be either sent to LabCorp (SC) or tested on site (EXP). On site testing of samples for EXP arm will occur in the same IPC room where rapid COVID-19 tests are tested. EXP panel results should be processed within 45 minutes to 1 hour but will be communicated to patient at COB (see below). Results will be communicated to both the patient and the health care provider as soon as possible, typically on the same day as enrollment. The research team will explain the results using a standarization script written by medical professionals. If patients have further questions, they will be referred to their healthcare provider. The usage of the RP EZ-2.1 Panel will guide the managemnet of providers in the following ways: more focused advice on time to isolate and/or quartine for patients, focused advice regarding infectivity, identifying the natural course of disease faster, guiding anti-biotic decisions for providers, and helping providers identify potential anti-viral therapy in a faster manner.

Patient data will be collected regarding demographics (Form D), comorbidities (Form D), nature of current symptoms (Form D), vaccination status (Form D), quality of life measures (Form E), vital signs at triage (Form F), CPT and ICD-10 codes (Form D), and travel history (Form D). This will be collected after the nasal swab is collected before the patient leaves the clinic. Patients will complete this form on a password protected iPad through secure REDCAP survey in a private, patient room. Patients will receive their results at the end of the day via follow up phone call by the research assistants (RAs) if randomized to the EXP group. If randomized to the SC group, patients will receive their results within 24-72 hours, dependent on turn around time at LabCorp. RAs will be providing results to both patients and providers. Providers can opt to complete a brief questionnaire (i.e., five minutes or less) regarding how their course of treatment was affected by the results. RAs will call patients to complete a brief satisfaction survey (15 minutes) with their results (if available) and uploaded results can be found in patient's electronic health record. Standardized scripts written by medical professionals will be used to provide diagnostic feedback for both patient groups via phone. Research assistants will provide diagnostic feedback to the providers in person for the EXP group. Clinician ordered testing (if any) can occur at any time and will be reported per usual protocol. If testing comes back positive for a bacterial/viral pathogen for EXP arm or SARS-COV-2 for SC arm, participants be referred to their health care provider if they want to seek further treatment or have questions about results. This is not inconsistent with the standard practices now happening at the IPCs. The study coordinator or trained research assistants will follow up with all enrolled patients at 7 business days to evaluate the course of symptoms, assess patient satisfaction, and to assess other relevant medical information.

ELIGIBILITY:
Inclusion Criteria:

* Age >7
* Clinically stable
* Must present with one symptom of respiratory illness (e.g., cough, sneezing, runny or stuffy nose, sore throat, headaches, muscle aches, trouble breathing, shortness of breath, and/or fever).

Exclusion Criteria:

* Patient is unable to provide informed consent
* Chronic symptoms (>14 days) or asymptomatic
* Unstable (or "too sick" to consent)
* Prisoner or ward of state
* Non-English speaker

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meltzer, MD, Principal Investigator — Clinical Research Director, Department of Emergency Medicine
Locations (2):
- United States (2):
  - GW Immediate & Primary Care - McPherson Square, Washington D.C., District of Columbia
  - GW Immediate & Primary Care - Rhode Island Ave, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided
We will consider per individual request, on case by case basis.

REFERENCES:
- [Background] Dugas AF, Valsamakis A, Atreya MR, Thind K, Alarcon Manchego P, Faisal A, Gaydos CA, Rothman RE. Clinical diagnosis of influenza in the ED. Am J Emerg Med. 2015 Jun;33(6):770-5. doi: 10.1016/j.ajem.2015.03.008. Epub 2015 Mar 12. PMID 25827595
- [Background] Beard K, Brendish N, Malachira A, Mills S, Chan C, Poole S, Clark T. Pragmatic multicentre randomised controlled trial evaluating the impact of a routine molecular point-of-care 'test-and-treat' strategy for influenza in adults hospitalised with acute respiratory illness (FluPOC): trial protocol. BMJ Open. 2019 Dec 17;9(12):e031674. doi: 10.1136/bmjopen-2019-031674. PMID 31852699
- [Background] Kim DK, Poudel B. Tools to detect influenza virus. Yonsei Med J. 2013 May 1;54(3):560-6. doi: 10.3349/ymj.2013.54.3.560. PMID 23549796
- [Background] Leber AL, Everhart K, Daly JA, Hopper A, Harrington A, Schreckenberger P, McKinley K, Jones M, Holmberg K, Kensinger B. Multicenter Evaluation of BioFire FilmArray Respiratory Panel 2 for Detection of Viruses and Bacteria in Nasopharyngeal Swab Samples. J Clin Microbiol. 2018 May 25;56(6):e01945-17. doi: 10.1128/JCM.01945-17. Print 2018 Jun. PMID 29593057
- [Background] Overview of influenza testing methods. Centers for Disease Control and Prevention. https://www.cdc.gov/flu/professionals/diagnosis/overview-testing-methods.htm. Published August 31, 2020. Accessed October 12, 2021.
- [Background] Poon SJ, Schuur JD, Mehrotra A. Trends in Visits to Acute Care Venues for Treatment of Low-Acuity Conditions in the United States From 2008 to 2015. JAMA Intern Med. 2018 Oct 1;178(10):1342-1349. doi: 10.1001/jamainternmed.2018.3205. PMID 30193357
- [Background] Weinick RM, Burns RM, Mehrotra A. Many emergency department visits could be managed at urgent care centers and retail clinics. Health Aff (Millwood). 2010 Sep;29(9):1630-6. doi: 10.1377/hlthaff.2009.0748. PMID 20820018

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Started | 205 | 155
Completed | 205 | 155
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care | Total
Number analyzed (Participants) | 205 | 155 | 360
Age, Customized [Median (Full Range); unit: years]
  Age (median age, years) | 34 [7 to 80] | 34 [7 to 89] | 34 [7 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 94 | 232
  Male | 67 | 61 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 10 | 29
  Not Hispanic or Latino | 184 | 145 | 329
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 7 | 20
  Native Hawaiian or Other Pacific Islander | 11 | 5 | 16
  Black or African American | 81 | 58 | 139
  White | 100 | 83 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Time to Receive Result
Description: Based on any results you have received from today's tests, are you satisfied in the time it has taken to communicate the results?
Time Frame: Day of enrollment
Measure: Number; unit: participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 183 | 125
participants
  Yes | 180 | 53
  No | 3 | 72

2. Secondary Outcome: Confidence in Testing
Description: Based on testing today, do you feel confident that you know what is causing your illness?
Time Frame: Day of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 183 | 125
Participants
  Yes | 111 | 37
  No | 43 | 57
  Unsure | 29 | 30
  Missing | 0 | 1

3. Secondary Outcome: Intention to Self Isolate
Description: Based on the testing you received today, are you planning to isolate from friends and family?
Time Frame: Day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 183 | 125
Participants
  Yes | 74 | 50
  No | 98 | 45
  Unsure | 9 | 27
  Not Applicable | 2 | 3

4. Secondary Outcome: Plan to Seek Care From Another Doctor or Healthcare Facility
Description: Will you seek out additional diagnostic testing or care from another doctor or healthcare facility?
Time Frame: Day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 183 | 125
Participants
  Yes | 30 | 17
  No | 134 | 80
  Unsure | 19 | 28

5. Secondary Outcome: Will Patient Plan for Work Absence
Description: Based on test results received today, will you plan to miss work?
Time Frame: Day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 183 | 125
Participants
  Yes | 62 | 60
  No | 78 | 42
  Not applicable | 43 | 23

6. Secondary Outcome: Did the Time to Receive Test Results Affect You and Prevent You From Doing Activities You Normally Would do?
Description: Did the time to receive test results affect you and prevent you from doing activities you normally would do?
Time Frame: Day 7 after enrollment
Measure: Number; unit: participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 156 | 124
participants
  Yes | 26 | 38
  No | 130 | 86

7. Secondary Outcome: I am Satisfied With the Time it Took to Receive the Test Results.
Time Frame: Day 7 after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 156 | 122
Participants
  Strongly agree/Agree | 145 | 73
  Neither agree or disagree | 7 | 16
  Strongly disagree/Disagree | 4 | 33

8. Secondary Outcome: Were Antibiotics Prescribed as Part of the IPC Visit for Respiratory Illness?
Description: Practitioner-Centered Results
Time Frame: Day of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 155 | 104
Participants
  Yes | 52 | 27
  No | 103 | 77

9. Secondary Outcome: Confidence in Patient's Cause of Illness
Description: How confident are you that you know what is causing your patient's illness?
Time Frame: Day of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
Number analyzed (Participants) | 155 | 104
Participants
  Less confident | 10 | 15
  No effect | 20 | 41
  More satisfied | 125 | 48

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events, and Other Adverse Events were monitored/assessed at Day 0 and Day 7
Arm/Group | BioFire® Respiratory Panel 2.1-EZ | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/155
Other Adverse Events (participants affected / at risk) | 0/205 | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT05467007/Prot_003.pdf
  • Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT05467007/SAP_001.pdf
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT05467007/ICF_002.pdf